CLINICAL TRIAL: NCT05681585
Title: Implementing Advanced Care Planning in the Routine Care for Acutely Admitted Patients in Geriatric Units: a Cluster Randomised Controlled Trial
Brief Title: Advanced Care Planning for the Severely Ill Home-dwelling Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo Metropolitan University (Other); Norwegian University of Science and Technology (Other); The Research Council of Norway (Other); Helse Sor-Ost (Other Government); Sykehuset Innlandet HF (Other); Vestre Viken Hospital Trust (Other); Ostfold Hospital Trust (Other); The Hospital of Vestfold (Other); Hospital of Southern Norway Trust (Other); University Hospital, Akershus (Other); Oslo University Hospital (Other); Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Reidar Pedersen, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NSD 805491
Record Dates: First submitted 2023-01-03; First posted 2023-01-12 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-12

CONDITIONS: Advance Care Planning
Keywords: Implementation science; Decision-making processes; Hospital; Geriatric; Next of kin; Clinical ethics; Qualitative methods; Cluster randomized clinical trial; Complex intervention; Health services for the aged; End of life
MeSH Terms: conditions — Death

STUDY DESIGN:
Intervention Model Description: The study is a cluster RCT, with a complex intervention containing implementation interventions and strategies, and a clinical intervention (ACP). Twelve clusters were recruited and stratified into two strata according to number of beds and randomized to intervention or control arms (allocation ratio of 1:1). The six hospital units in the intervention arm will receive a comprehensive implementation support program, whereas the control units receive no support in the intervention period.
  A similar number of patients, relatives and attending clinician will be recruited from both arms in triads for the quantitative sub-study. Data for each patient will be supplemented by health record and register data. Patients, relatives, staff and implementation teams will be recruited from the intervention units to qualitative interviews. All health personnel in the participating units will be recruited to answer a questionnaire twice. We will also interview key stakeholders in a wider context.
Masking Description: No masking Patients and next-of-kin will not be informed about the hospital unit's allocation status. However, they may deduce this from the kind of intervention they receive. It's impossible to blind the care providers and for practical reasons we won't be able to blind the investigators or the outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Other): Clusters (medical/geriatric hospital units) in the intervention arm receives a comprehensive implementation support program during the trial period.
  Interventions: Other: Implementation support program
- Control arm (No Intervention): Clusters (medical/geriatric hospital units) in the control arm receives no implementation support program during the trial period.
  These units will receive the implementation support program after the trial period.

INTERVENTIONS:
Other: Implementation support program — The intervention consists of:
  I Implementation strategies:
  1.1 Ensuring leadership commitment 1.2 Responsive evaluation 1.3 Whole ward approach 1.4 Train the trainer model 1.5 Sustainability after the study
  II Implementation interventions 2.1 Implementation team 2.2 ACP coordinator 2.3 Training and supervision: Kick-off, training of resource persons and health care personnel including practical exercises, network conferences 2.4 Toolkit and shared resources: ACP guideline, teaching material, information leaflets, documentation templates etc. 2.5 Structured fidelity measurements of the implementation level of a) the implementation interventions and b) the clinical intervention, with tailored feedback and supervision
  III Clinical intervention: Advance Care Planning 3.1 Routine information and invitation to Advance Care Planning to all eligible patients 3.2 Written information to patients and relatives 3.3 Documentation and collaboration with other health care levels
  Arms: Intervention arm

SUMMARY:
This study will develop and evaluate a complex intervention to implement advance care planning for severely ill home-dwelling elderly acutely admitted to hospital, by using a cluster randomized design.

Twelve Norwegian acute geriatric hospital units will participate in the main study, each as one cluster. Of the twelve clusters, half will receive implementation support and training immediately, and the other half will receive similar support after the intervention period. The study includes 1) assessment of implementation outcomes (fidelity) in the participating units,2) health service and clinical outcomes including a) questionnaires to all staff in the units before and after the implementation period, questionnaires to attending clinicians and qualitative interviews with health personnel and local unit leaders b) questionnaires to patients and their relatives, patients records and data from central health registers and qualitative interviews with patients and relatives. Furthermore we will assess barriers and facilitators for advance care planning in 1) a wider health service context, and 2) at the national, regional and municipal level, and do economic analyses.

DETAILED DESCRIPTION:
Background:

Severely ill elderly patients and their relatives are often poorly involved in treatment and care decisions. Advance care planning is a well-documented tool to comply with the ethical and legal imperative to involve both the patient and their next of kin in the planning of current and future treatment and care. The overall aim of this project is to improve health services, user involvement and quality of life for severely ill elderly people living at home, and their relatives, in an efficient, sustainable and coordinated way, through better implementation of Advance care planning (ACP).

Setting: Twelve hospital wards providing care to acutely admitted elderly home-dwelling patients, either pure geriatric units or mixed units with specialists in geriatric medicine.

Research questions:

1. What is the current level of implementation of ACP for home-dwelling elderly patients with severe somatic disease in the participating clinical units?
2. What are the most important facilitators and barriers among all relevant stakeholders - to implementing ACP at the a) clinical, b) health care service- and c) national, regional and municipal level?
3. What are the most important moral dilemmas and conflicting interests related to ACP, and how can these be resolved?
4. What are the benefits and disadvantages with the implementation support and ACP experienced by the patients, among next of kin, health personnel and implementation teams?
5. Does the implementation support program - compared to no such support - improve a) the implementation of ACP (fidelity), b) quality of communication and decision-making for patients and relatives when approaching the end of life, and c) congruence between the patient's preferences for information and involvement and the attending clinician's perceptions of the same, and other relevant outcomes for patients, relatives, and the attending clinicians?
6. Is the implementation support program associated with changes in health personnel's perceptions, attitudes, self-efficacy, confidence in, and experiences in relation to information giving and involvement of patients and relatives?
7. Is higher level of implementation (fidelity) of ACP associated with improved outcomes for patients, relatives, the staff and the services?
8. Is the implementation support program for ACP a cost-effective intervention?

Hypotheses:

1. The current level of implementation of ACP for home-dwelling elderly patients with severe somatic disease in participating clinical units is low.
2. There are important facilitators for and barriers to implementing ACP among all stakeholders at the a) clinical, b) health care service- and c) national and other higher levels.
3. There are important moral dilemmas and conflicting interests related to ACP, and they can be dealt with through systematic approaches and ethics reflection.
4. Patients, among next of kin, health personnel and implementation teams experience both benefits and disadvantages with the implementation support and ACP.
5. The implementation support program - compared to no such support - will improve a) improve the implementation of ACP (fidelity), b) quality of communication and decision-making for patients and relatives when approaching the end of life, and c) congruence between the patient's preferences for information and involvement and the attending clinician's perceptions of the same, and other relevant outcomes for patients, relatives, and the attending clinicians.
6. The implementation support program is associated with changes in health personnel's perceptions, attitudes, self-efficacy, confidence in, and experiences in relation to information giving and involvement of patients and relatives
7. Higher level of implementation (fidelity) of ACP is associated with improved outcomes for patients, relatives, the staff and the services
8. Outcomes for patients, relatives and the public health- and welfare services justify the costs of the implementation support program and of ACP in routine care.

ELIGIBILITY:
Inclusion and exclusion criteria for patients and relatives the quantitative and triadic sub-study:

Inclusion criteria for patients:

* Home-dwelling
* 70 years or older
* Acutely admitted to the participating unit
* Sufficient language proficiency in Norwegian to answer the questionnaire
* Clinical frailty score of 4 or more
* The physician responsible for the patient's medical care answers "no" to "Surprise question" from Gold Standards Framework proactive identification guidance
* Both patient and a close relative (preferably the closest relative) would participate in ACP together if offered
* Both patient and the close relative consent to participate in the research project

Exclusion criteria for patients:

* The patient is not competent to consent to research participation
* The patient is expected to die within 24 hours
* The patient has participated in ACP prior to the current hospital admission
* In the intervention arm

  * ACP is not conducted with patient, next of kin and physician before hospital discharge
  * The clinician that participated in the ACP conversation has not consented to research participation
* In the control arm

  * The patient would not have been able to participate in ACP during hospitalization
  * An attending clinician has not consented to research participation

Inclusion criteria for relatives:

* A close relative of a patient who fulfill all inclusion criteria and no exclusion criteria; and who would be willing to participate in ACP together with the patient if offered
* 18 years or older
* Sufficient language proficiency in Norwegian to answer the questionnaire
* Both patient and the close relative consent to participate in the research project

Exclusion criteria for relatives:

* The relative is not competent to consent to research participation
* In the intervention arm

  * ACP is not carried out with the patient, next of kin and attending clinician before hospital discharge
* In the control arm

  * The relative would not have been able to participate in ACP during hospitalization

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Implementation outcome study: Fidelity to the intervention model - Advanced Care Planning | Baseline, 9 and 18 months in the intervention arm. Baseline and 18 months in the control arm.
  Change in fidelity (sum score) measured by the fidelity scale for Advanced Care Planning. Rated from 1 (low) to 5 (high).
Clinical effectiveness study 1: Patient-reported outcome | During the intervention period (10-18 months after the start of the implementation support)
  Quality of communication and decision-making when the patient is approaching the end of life. 4 items, scale 0-9.
Clinical effectiveness study 2: Relative-reported outcome | During the intervention period (10-18 months after the start of the implementation support)
  Quality of communication and decision-making for the patient and the next-of-kin when approaching the end of life. 4 items, rated 0-9.
Clinical effectiveness study 3: Clinician outcome | During the intervention period (10-18 months after the start of the implementation support)
  Congruence between the patient's preferences for information and involvement and the attending clinician's perceptions of the same, 4 items, scales: 0-9, 0-2, 0-9, 7 alternative answers, respectively

SECONDARY OUTCOMES:
Implementation outcome study: Fidelity to the intervention model - Advanced Care Planning 1 | Baseline, 9 and 18 months in the intervention arm. Baseline and 18 months in the control arm.
  Change in fidelity subscale - Organizational implementation - measured by the fidelity scale for Advanced Care Planning. Rated from 1 (low) to 5 (high).
Implementation outcome study: Fidelity to the intervention model - Advanced Care Planning 2 | Baseline, 9 and 18 months in the intervention arm. Baseline and 18 months in the control arm.
  Change in fidelity subscale - Quality of ACP - measured by the fidelity scale for Advanced Care Planning. Rated from 1 (low) to 5 (high).
Implementation outcome study: Fidelity to the intervention model - Advanced Care Planning 3 | Baseline, 9 and 18 months in the intervention arm. Baseline and 18 months in the control arm.
  Change in fidelity subscale - Penetration - measured by the fidelity scale for Advanced Care Planning. Rated from 1 (low) to 5 (high).
Clinical effectiveness study 1: Patient-reported seondary outcome 1 | During the intervention period (10-18 months after the start of the implementation support)
  Communication about preferences for information and involvement, providers' current compliance with these preferences, and trust in future compliance. 5 items, rated 0-9.
Clinical effectiveness study 1: Patient-reported seondary outcome 2 | During the intervention period (10-18 months after the start of the implementation support)
  Satisfaction with information and involvement concerning health care provided during admittance and that will be provided after discharge, and with information about the patient's state of health, discharge, prognosis and future health care needs. 10 items, rated 0-9
Clinical effectiveness study 1: Patient-reported seondary outcome 3 | During the intervention period (10-18 months after the start of the implementation support)
  Self-efficacy in communicating with next-of-kin and health care professionals about future deterioration, preferences for life-prolonging treatment in such a situation, and health care when approaching the end of life. 9 items, rated 0-3
Clinical effectiveness study 1: Patient-reported seondary outcome 4 | During the intervention period (10-18 months after the start of the implementation support)
  Problem causing admittance solved, satisfaction with arrival, stay, and discharge at the hospital, and trust in necessary health care in the future. 5 items, rated 0-9
Clinical effectiveness study 1: Patient-reported seondary outcome 5 | During the intervention period (10-18 months after the start of the implementation support)
  Concrete preferences for information and who should participate in important decisions about health care, and assessment of the amount of information given. 4 items, scales: 0-9, 0-2, 0-9, 7 alternative answers, respectively
Clinical effectiveness study 1: Patient-reported seondary outcome 6 | During the intervention period (10-18 months after the start of the implementation support)
  General life satisfaction (ref. OECD. (2013). OECD guidelines on measuring subjective well-being). 1 item, rated 0-10.
Clinical effectiveness study 1: Patient registry data 1 - Number of hospital admissions | From 18 months before to 18 months after inclusion (or until death)
  Retrieved from national registries
Clinical effectiveness study 1: Patient registry data 2 - Other use of health care services and use of medication | From 18 months before to 18 months after inclusion (or until death)
  Retrieved from national registries
Clinical effectiveness study 1: Patient registry data 3 - Time before death (for patients dying before 18 months after inclusion) | From inclusion to 18 months after inclusion
  Retrieved from national registries
Clinical effectiveness study 1: Patient health records data | From 18 months before to 18 months after inclusion (or until death)
  Documentation concerning ACP and other similar conversations, palliative care plan, the patient's life stance or religious beliefs, and life prolonging treatment and palliative care given and any decisions to limit such treatment or care, and similarly for hospital admittance.
Clinical effectiveness study 2: Relative-reported seondary outcome 1 | During the intervention period (10-18 months after the start of the implementation support)
  Satisfaction with information and involvement concerning the patient's health care provided during admittance and that will be provided after discharge, with information about the patient's state of health, discharge, prognosis, future health care needs, and with the providers' understanding of the next-of-kin's situation. 11 items, rated 0-9
Clinical effectiveness study 2: Relative-reported seondary outcome 2 | During the intervention period (10-18 months after the start of the implementation support)
  Self-efficacy in communicating with the patient and health care professionals about future deterioration, the patient's preferences for life-prolonging treatment in such a situation, and health care when the patient is approaching the end of life. 9 items, rated 0-3.
Clinical effectiveness study 2: Relative-reported seondary outcome 3 | During the intervention period (10-18 months after the start of the implementation support)
  Problem causing admittance solved, satisfaction with arrival, stay, and discharge at the hospital, trust in necessary health care for the patient in the future, and make sure that the patient receives needed health care in the time to come. 6 items, ratet 0-9.
Clinical effectiveness study 2: Relative-reported seondary outcome 4 | During the intervention period (10-18 months after the start of the implementation support)
  Next-of-kin's concrete preferences for information and assessment of the amount of information given, the patient's preference for information and who should participate in important decisions about health care. 4 items, scales: 0-9, 0-2, 0-9, 7 alternative answers, respectively
Clinical effectiveness study 2: Relative-reported seondary outcome 5 | During the intervention period (10-18 months after the start of the implementation support)
  Next-of-kin's tasks and burdens. 7 items with various scales/response alternatives.
Clinical effectiveness study 2: Relative-reported seondary outcome 6 | During the intervention period (10-18 months after the start of the implementation support)
  Informal carer's care-related quality of life (ref. CarerQoL-7D (Brouwer et al. 2006)). 7 items, rated 0-2
Clinical effectiveness study 2: Relative-reported seondary outcome 7 | During the intervention period (10-18 months after the start of the implementation support)
  General life satisfaction (ref. OECD. (2013). OECD guidelines on measuring subjective well-being). 1 item, rated 0-10.
Clinical effectiveness study 3: Clinician secondary outcome 1 | During the intervention period (10-18 months after the start of the implementation support)
  Self-confidence in matching involvement of patient and next-of-kin and future decision-making to patient's preferences. 4 items, rated 0-10
Clinical effectiveness study 3: Clinician secondary outcome 2 | During the intervention period (10-18 months after the start of the implementation support)
  Self-efficacy in communicating about future deterioration, preferences for life-prolonging treatment in such a situation, for future care (at home or in a nursing home), and for health care when approaching the end of life, with the patient, next-of-kin, and other providers. 16 items, rated 0-3.
Clinical effectiveness study 4: All staff - 1 | Baseline and 18 months in both intervention and control arm
  Patients' and relatives' preferences for information and involvement. 7 questions.
Clinical effectiveness study 4: All staff - 2 | Baseline and 18 months in both intervention and control arm
  Whether information, involvement and health care provided is concordant with the patients' and relatives' preferences, and reasons for discordance. 9 questions.
Clinical effectiveness study 4: All staff - 3 | Baseline and 18 months in both intervention and control arm
  Decision making authority - clinical realities and ideals. 16 questions.
Clinical effectiveness study 4: All staff - 4 | Baseline and 18 months in both intervention and control arm
  Self-efficacy in ACP-relevant information and involvement tasks.17 questions.
Clinical effectiveness study 4: All staff - 5 | Baseline and 18 months in both intervention and control arm.
  Self-confidence in ACP-relevant information and involvement tasks. 7 questions.
Economic sub-study: Increased costs related to implementing and practicing ACP | Measured before baseline and then throughout the implementation period (0-18 months).
  Increased costs related to implementing and practicing ACP in the clinical units in the intervention arm. Compared to normal costs before baseline. Differences in costs will be compared to the primary outcomes (differences measured as percentage point) and selected secondary outcomes.

OTHER OUTCOMES:
Clinical effectiveness study 1: Clinical data about the patient from participating/attending clinician | During the intervention period (10-18 months after the start of the implementation support)
  We ask the participant clinician (clinical effectiveness study 3) to report key clinical information about the patient. 14 items in the intervention units, and 15 items in the control units, with various scales/response alternatives, including free text answers (e.g. main diagnosis).

CONTACTS AND LOCATIONS:
Overall Officials: Reidar Pedersen, PhD, Principal Investigator — Professor, Centre for medical ethics, University of Oslo
Locations (12):
- Norway (12):
  - Vestre Viken Hospital Trust, Bærum, Oslo, Bærum kommune
  - Hospital of Southern Norway, Arendal, Arendal
  - Vestre Viken Hospital Trust, Drammen, Drammen
  - Innlandet Hospital Trust, Elverum, Elverum
  - Innlandet Hospital Trust, Gjøvik, Gjøvik
  - Vestre Viken Hospital Trust, Kongsberg, Kongsberg
  - Hospital of Southern Norway, Kristiansand, Kristiansand
  - Akershus University Hospital, Lørenskog
  - Diakonhjemmet Hospital, Oslo
  - Oslo University Hospital, Oslo
  - Østfold Hospital Trust, Sarpsborg
  - Vestfold Hospital Trust, Tønsberg

IPD SHARING:
Plan to Share IPD: No
Anonymized data and documents from all sub-studies can be made available to other researchers upon request after project end, in the period April 19 2032 - April 19 2037.
  What types of analyses and with what mechanism data will be made available will be planned if relevant.

REFERENCES:
- [Background] Detering KM, Hancock AD, Reade MC, Silvester W. The impact of advance care planning on end of life care in elderly patients: randomised controlled trial. BMJ. 2010 Mar 23;340:c1345. doi: 10.1136/bmj.c1345. PMID 20332506
- [Background] Molloy DW, Guyatt GH, Russo R, Goeree R, O'Brien BJ, Bedard M, Willan A, Watson J, Patterson C, Harrison C, Standish T, Strang D, Darzins PJ, Smith S, Dubois S. Systematic implementation of an advance directive program in nursing homes: a randomized controlled trial. JAMA. 2000 Mar 15;283(11):1437-44. doi: 10.1001/jama.283.11.1437. PMID 10732933
- [Background] Lund S, Richardson A, May C. Barriers to advance care planning at the end of life: an explanatory systematic review of implementation studies. PLoS One. 2015 Feb 13;10(2):e0116629. doi: 10.1371/journal.pone.0116629. eCollection 2015. PMID 25679395
- [Background] Rietjens JAC, Sudore RL, Connolly M, van Delden JJ, Drickamer MA, Droger M, van der Heide A, Heyland DK, Houttekier D, Janssen DJA, Orsi L, Payne S, Seymour J, Jox RJ, Korfage IJ; European Association for Palliative Care. Definition and recommendations for advance care planning: an international consensus supported by the European Association for Palliative Care. Lancet Oncol. 2017 Sep;18(9):e543-e551. doi: 10.1016/S1470-2045(17)30582-X. PMID 28884703
- [Background] Weathers E, O'Caoimh R, Cornally N, Fitzgerald C, Kearns T, Coffey A, Daly E, O'Sullivan R, McGlade C, Molloy DW. Advance care planning: A systematic review of randomised controlled trials conducted with older adults. Maturitas. 2016 Sep;91:101-9. doi: 10.1016/j.maturitas.2016.06.016. Epub 2016 Jun 23. PMID 27451328
- [Background] Brinkman-Stoppelenburg A, Rietjens JA, van der Heide A. The effects of advance care planning on end-of-life care: a systematic review. Palliat Med. 2014 Sep;28(8):1000-25. doi: 10.1177/0269216314526272. Epub 2014 Mar 20. PMID 24651708
- [Background] Bernacki RE, Block SD; American College of Physicians High Value Care Task Force. Communication about serious illness care goals: a review and synthesis of best practices. JAMA Intern Med. 2014 Dec;174(12):1994-2003. doi: 10.1001/jamainternmed.2014.5271. PMID 25330167
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Derived] Broderud L, Romoren M, Hermansen KB, Saevareid TJL, Thoresen L, Pedersen R. Barriers and facilitators in implementing advance care planning for frail older patients acutely admitted to geriatric hospital units: a nested qualitative study. Front Health Serv. 2025 Dec 17;5:1646541. doi: 10.3389/frhs.2025.1646541. eCollection 2025. PMID 41479948
- [Derived] Westbye SF, Romoren M, Ahmed M, Hermansen KB, Broderud L, Wahl AK, Saevareid TJL, Thoresen L, Pedersen R. Measuring the level of implementation of advance care planning - a fidelity-based cross-sectional study. Front Health Serv. 2025 Oct 29;5:1629242. doi: 10.3389/frhs.2025.1629242. eCollection 2025. PMID 41234374
- [Derived] Romoren M, Hermansen KB, Saevareid TJL, Broderud L, Westbye SF, Wahl AK, Thoresen L, Rostoft S, Forde R, Ahmed M, Aas E, Midtbust MH, Pedersen R. Implementation of advance care planning in the routine care for acutely admitted patients in geriatric units: protocol for a cluster randomized controlled trial. BMC Health Serv Res. 2024 Feb 19;24(1):220. doi: 10.1186/s12913-024-10666-0. PMID 38374100
- See also: Gold Standards Framework. Advance care planning 2019 — http://www.goldstandardsframework.org.uk/advance-care-planning